CLINICAL TRIAL: NCT03017872
Title: A Phase IIIB/IV Randomised Open-label Trial Comparing Dolutegravir With Pharmaco-enhanced Darunavir Versus Dolutegravir With Predetermined Nucleosides Versus Recommended Standard of Care ART Regimens in Patients With HIV-1 Infection Failing First Line Therapy.
Brief Title: Dolutegravir and Darunavir Evaluation in Adults Failing Therapy
Acronym: D²EFT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kirby Institute (Other Government)
Collaborators: UNITAID (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Health and Medical Research Council, Australia (Other); ViiV Healthcare (Industry); Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2EFT; 18Q065 (Other Grant/Funding Number: NIAID via Leidos); 19Q120 (Other Grant/Funding Number: NIAID via Leidos)
Record Dates: First submitted 2017-01-02; First posted 2017-01-11 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: HIV, second-line
MeSH Terms: conditions — HIV Infections | interventions — Nucleosides; dolutegravir; Darunavir; Ritonavir

STUDY DESIGN:
Intervention Model Description: A third arm has been incorporated using a multi-arm, multi-stage (MAMS) design. This design allows for the 2-arm study (DTG+DRV/r vs DRV/r+2NRTI) to continue accrual while preparation of the new arm (DTG+2NRTI) is begun in parallel. Once that arm is ready, accrual to it begins and the study switches to the second stage. All participants accrued to Arm 1 and 2 throughout the trial are contemporaneous and can be compared, while the subjects accrued to Arm 3 are compared only to their contemporaries in Arms 1 and 2. The size of Arm 3 is sufficient to allow adequate power comparisons, and stage effects are minimized while non-contemporaneous control data are not required.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard of Care (SoC) arm (Active Comparator): 2 x NRTIs + darunavir/ritonavir 800mg/100mg po od
  Interventions: Drug: NRTIs; Drug: Darunavir; Drug: Ritonavir
- Dolutegravir arm (Experimental): Dolutegravir 50mg + darunavir/ritonavir 800mg/100mg po od
  Interventions: Drug: Dolutegravir; Drug: Darunavir; Drug: Ritonavir
- Dolutegravir 2NRTI arm (D2N) (Experimental): Dolutegravir 50mg + 2 x NRTIs (tenofovir plus emtricitabine or lamivudine)
  Interventions: Drug: NRTIs; Drug: Dolutegravir

INTERVENTIONS:
Drug: NRTIs — In SOC arm, choice of NRTIs determined by clinician, guided by either genotypic resistance testing or use of a protocol-specified algorithm for N(t)RTI selection.
  In D2N arm, NRTIs are predetermined.
  Other Names: Nucleoside/Nucleotide Reverse Transcription Inhibitors
  Arms: Dolutegravir 2NRTI arm (D2N); Standard of Care (SoC) arm
Drug: Dolutegravir — 50mg tablet by mouth once daily for 96 weeks.
  Other Names: Tivicay
  Arms: Dolutegravir 2NRTI arm (D2N); Dolutegravir arm
Drug: Darunavir — 800mg tablet by mouth once daily for 96 weeks.
  Other Names: Prezista
  Arms: Dolutegravir arm; Standard of Care (SoC) arm
Drug: Ritonavir — 100mg tablet by mouth once daily for 96 weeks.
  Other Names: Norvir
  Arms: Dolutegravir arm; Standard of Care (SoC) arm

SUMMARY:
D²EFT is a randomised, open-label study in HIV-1 infected patients failing first-line antiretroviral therapy (ART). The study compares 2 regimens of second-line ART (dolutegravir and darunavir pharmaco-enhanced with ritonavir and dolutegravir and 2 prespecified NRTIs) with the WHO recommended regimen of 2NRTIs plus a ritonavir-boosted PI (Standard of Care (SOC)). 1,010 participants from 14 predominantly low-middle income countries will be followed for 96 weeks with the primary endpoint at week 48. The design is based on the hypothesis that one or both of the new regimens will be non-inferior to SOC in terms of virologic control while being easier to take, economically viable and affording simplification of treatment programs.

DETAILED DESCRIPTION:
Consenting participants will be screened and within 45 days randomly allocated to receive either dolutegravir and darunavir/ritonavir, dolutegravir and 2 prespecified NRTIs or the SOC regimen. Participants will be seen four weeks after their randomisation (week 0) visit and then at weeks 12, 24, 48 and 96. Consenting participants will have storage samples collected and cryopreserved at their week 0, 48 & 96 visits. This repository will be used in future for central baseline resistance testing, pharmacogenomic testing (separate consent required) and has inherent value for later studies of HIV pathogenesis. A 1-time PK sample will be collected at week four for future testing and any participants failing therapy at 24 weeks will have a plasma sample stored for future genotypic resistance testing.

A number of secondary outcomes will be considered in order to compare the performance of the two study treatment regimens. Secondary analyses will focus on virological, immunological, safety, antiretroviral treatment change and medication adherence. A comparison of costs and estimates of cost-effectiveness for the randomised comparison will be a critical component of this study. ART costs will be assessed across study arms. Health-care utilisation will be self-reported and then used to estimate costs. Safety data, viral loads and quality of life data will also be analysed.

The open label nature of the study allows routine care to be undertaken and the use of objective endpoints limit potential bias. The study has well defined and integrated clinical data collection and patient management systems that have been shown to be effective in a wide range of clinical settings.

The choice of NRTIs in the SoC regimen is based on clinical judgement and may be guided by resistance testing if locally available, while those used with dolutegravir are predetermined (tenofovir and lamivudine or emtricitabine). The NRTIs are not provided via the study. At the end of 96 weeks (completion of the protocol) study drug can be offered to all participants for a further 48 weeks as informed by the 48-week study results and clinical judgement. After 144 weeks study drug will no longer be available and composition of the participant's post-study regimen will be the clinician's decision.'

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive by licensed diagnostic test
2. Aged ≥16 years of age (or minimum age as determined by local regulations or as legal requirements dictate)
3. Failed first-line non-nucleoside reverse transcriptase inhibitor (NNRTI) + 2N(t)RTI combination therapy according to virological criteria, defined as at least two consecutive (≥7 days apart) pVL results >500 copies/mL after a minimum period of exposure to continuous NNRTI + 2N(t)RTI first-line therapy of 24 weeks (only the second pVL result needs to be within 45 days of randomisation)
4. For women of child-bearing potential, willingness to use appropriate contraception
5. Able to provide written informed consent

Exclusion Criteria:

1. The following laboratory variables:

   1. absolute neutrophil count (ANC) <500 cells/µL
   2. haemoglobin <7.0 g/dL
   3. platelet count <50,000 cells/µL
   4. AST and/or ALT ≥5xULN OR ALT ≥3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin)
2. Change in antiretroviral therapy within 12 weeks prior to randomisation
3. Prior exposure to HIV protease inhibitors and/or HIV integrase inhibitors
4. Patients with chronic viral hepatitis B infection defined by positive serum hepatitis B surface antigen
5. Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy (INR >2.3), hypoalbuminemia (serum albumin <2.8g/dL), esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
6. Anticipated need for Hepatitis C virus (HCV) therapy during the study
7. Subject has creatinine clearance of <50 mL/min via CKD-EPI equation
8. Current use of rifabutin or rifampicin
9. Use of any contraindicated medications (as specified by product information sheets)
10. Intercurrent illness requiring hospitalization
11. An active opportunistic disease not under adequate control in the opinion of the investigator
12. Pregnant or nursing mothers
13. Patients with current alcohol or illicit substance use that in the opinion of the investigator might adversely affect participation in the study
14. Patients deemed unlikely by the investigator to be able to remain in follow-up for the protocol-defined period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 831 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants in each arm whose plasma viral load is <50 copies/mL at 48 weeks by intention to treat. | At 48 weeks

SECONDARY OUTCOMES:
Proportion with plasma viral load <200 copies/mL | At 48 and 96 weeks
Proportion with plasma viral load <50 copies/mL where those stopping randomised therapy for any reason are classified as plasma viral load >50 copies/mL | At 48 and 96 weeks
Mean change in CD4+ cell count from baseline | At 48 and 96 weeks
Mean/median changes from baseline in fasted lipids (Total cholesterol, LDL-c, HDL-c, and triglycerides) | At 48 and 96 weeks
Total number of participants with any serious adverse events (SAEs), and the cumulative incidence of SAEs | At 48 and 96 weeks
Total number of opportunistic diseases (AIDS events), deaths and serious non-AIDS defining events and the cumulative incidence of these | At 48 and 96 weeks
Adverse events associated with cessation of randomly assigned therapy | At 48 and 96 weeks
Categorisation of neuropsychological adverse events | At 48 and 96 weeks
Proportion who stopped randomised therapy by reason for stopping | At 48 and 96 weeks
Patterns of genotypic HIV resistance associated with virological failure | At 48 and 96 weeks
Adherence assessment using participant 7-day recall self-report questionnaire | At week 4
Quality of life and anxiety & depression assessed by participant questionnaire | At 48 and 96 weeks
Health care utilisation assessed by participant questionnaire | At 48 and 96 weeks
Cost of care assessment | At 48 and 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail Matthews, MD, Principal Investigator — Kirby Institute
Locations (28):
- Argentina (4):
  - Hospital Dr Diego Paroissien, Isidro Casanova, Buenos Aires
  - Hospital G de Agudos JM Ramos Mejia, Buenos Aires, Buenos Aires F.D.
  - CAICI, Rosario, Santa Fe Province
  - Hospital Interzonal de Agudos San Juan de Dios, La Plata
- Laboratório de Pesquisa Clinica Em Hiv/Aids - Instituto Nacional de Infectologia - Fiocruz, Rio de Janeiro, Brazil
- Hospital San Borja-Arriaran, Santiago, Chile
- ASISTENCIA Cientifica De Alta Complejidad S.A.S., Bogotá, Colombia
- Centre de traitementambulatoire de Donka ( Hopital de jour), Conakry, Guinea
- CART CRS, VHS Hospital, Chennai, Tamil Nadu, India
- Indonesia (4):
  - Dr. Cipto Mangunkusumo Hospital, Jakarta
  - RSUP Dr. Wahidin Sudirohusodo, Makassar
  - Dr. Soetomo Hospital, Surabaya
  - Dr Sardjito Hospital, Yogyakarta
- Malaysia (2):
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - University of Malaya Medical Centre, Kuala Lumpur
- University of Sciences, Techniques and Technologies of Mali, University Clinical Research Center (UCRC), Bamako, Mali
- Mexico (3):
  - Morales Vargas Centro de Investigacion SC, León, Guanajuato
  - Hospital Civil de Guadalajara, Guadalajara, Jalisco
  - Instituto Nacional de Ciencias Medicas y Nutriciòn Salvador Zubiran, Mexico City
- Institute of Human Virology, Nigeria (IHVN), Abuja, Nigeria
- South Africa (3):
  - Desmond Tutu HIV Foundation, Cape Town
  - Clinical HIV Research Unit (CHRU), Wits Health Consotium (Pty) Ltd, Johannesburg
  - Perinatal HIV Research Unit (PHRU), Chris Hani Baragwanath Hospital, Soweto
- Thailand (4):
  - HIV-NAT (The HIV Netherlands Australia Thailand Research Collaboration), Thai Red Cross AIDS Research Centre, Bangkok
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D2EFT Study Group. Dolutegravir plus boosted darunavir versus recommended standard-of-care antiretroviral regimens in people with HIV-1 for whom recommended first-line non-nucleoside reverse transcriptase inhibitor therapy has failed (D2EFT): an open-label, randomised, phase 3b/4 trial. Lancet HIV. 2024 Jul;11(7):e436-e448. doi: 10.1016/S2352-3018(24)00089-4. Epub 2024 May 21. PMID 38788744
- [Derived] Nyein PP, Petoumenos K, Borok M, Eriobu N, Kumarasamy N, Avihingsanon A, Azwa I, Dao S, Cisse M, Dharan NJ, Hanson J, Matthews GV. Associations Between Antiretroviral Regimen and Changes in Blood Pressure: Results From the D2EFT Study. Clin Infect Dis. 2025 Feb 5;80(1):160-163. doi: 10.1093/cid/ciae256. PMID 38721980